CLINICAL TRIAL: NCT02711527
Title: Activation on Left Dorsolateral Prefrontal Cortex LDPC With Different Acupoint-Combinations for Depression: An fNIRS Study
Brief Title: Activation on LDPC Cortex With Different Acupoints: An fNIRS Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wu Junmei, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW16-008
Record Dates: First submitted 2016-02-23; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupunture group A (Active Comparator): The subjects will receive acupuncture treatment twice weekly for 3 weeks (6 treatments in total) Subjects in Group A will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation" , all needles will be retained for 30 minutes.
  Interventions: Other: Acupunture group A
- Acupunture group B (Active Comparator): The subjects will receive acupuncture treatment twice weekly for 3 weeks (6 treatments in total). Subjects in Group B will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation" and "Tonifying the heart and the spleen"and "Invigorating the Yang Qi", all needles will be retained for 30 minutes.
  Interventions: Other: Acupunture group B

INTERVENTIONS:
Other: Acupunture group A — Subjects in Group A will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation", all needles will be retained for 30 minutes. Acupoint combination: Taichong太衝 (LR 3), Ligou蠡沟 (LR 5), Zhongdu 中都(LR6), Xiguan膝關 (LR 7), Ququan曲泉 (LR 8), Zhangmen章門(LR13), Qimen期門 (LR14).
  Arms: Acupunture group A
Other: Acupunture group B — Subjects in Group B will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation" and "Tonifying the heart and the spleen"and "Invigorating the Yang Qi", all needles will be retained for 30 minutes. Acupoint combination: Taichong太衝 (LR 3), , Sanyinjiao 三陰交 (SP 6), Xuanzhong懸鐘 (GB 39), Shenmen 神門 (HT 7), Zusanli 足三里(ST 36), Baihui 百會(DU 20), Shenting神庭(DU24), Qihai 氣海(RN6), Guanyuan 關元(RN4). Teding Diancibo Pu (abbreviation: TDP) "特定電磁波譜" will be applied to Group B immediately after the needle insertion.
  Arms: Acupunture group B

SUMMARY:
This is a randomized, open-labelled study to study the effect of the different acupoints combination under TCM treatment principles by fNIRS.

The investigator aim to recruited 36 depression subjects and go through 6 acupuncture treatment sessions in 3 weeks. They will be divided into 2 groups by randomization. (Group A n=18, Group B n=18) The participants will receive 2 acupuncture session per week for 3 consecutively weeks. In each treatment session, all subjects in both groups will receive the same amount of needle insertion ( total 14 needles) , all needles will be retained for 30 minutes. The whole treatment will last for around 45 minutes. No sedation will be conducted.

Subjects in Group A will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation", all needles will be retained for 30 minutes. Acupoint combination: Taichong太衝 (LR 3), Ligou蠡沟 (LR 5), Zhongdu 中都(LR6), Xiguan膝關 (LR 7), Ququan曲泉 (LR 8), Zhangmen章門(LR13), Qimen期門 (LR14).

Subjects in Group B will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation" and "Tonifying the heart and the spleen"and "Invigorating the Yang Qi", all needles will be retained for 30 minutes. Acupoint combination: Taichong太衝 (LR 3), , Sanyinjiao 三陰交 (SP 6), Xuanzhong懸鐘 (GB 39), Shenmen 神門 (HT 7), Zusanli 足三里(ST 36), Baihui 百會(DU 20), Shenting神庭(DU24), Qihai 氣海(RN6), Guanyuan 關元(RN4). Teding Diancibo Pu (abbreviation: TDP) "特定電磁波譜" will be applied to Group B immediately after the needle insertion. This TDP device is a infra-red heat lamp which is commonly used by acupuncturists and Chinese Medicine Practitioner as a therapeutic substitute for moxibustion. The procedure will be lasted for 30 minutes in 30-40 cm above the specified acupoint Qihai 氣海(RN6) and Guanyuan 關元(RN4).

DETAILED DESCRIPTION:
This is a randomized, open-labelled study to study the effect of the different acupoints combination under TCM treatment principles by fNIRS.

The investigator aim to recruited 36 depression subjects and go through 6 acupuncture treatment sessions in 3 weeks. The subjects will be asked to visit the clinic for 7 times. The depression subjects will be recruited from Queen Mary Hospital, The Mental Health Association of Hong Kong (Kwun Tong center) and the community. Basic personal information, depression medical history, level of education etc will be collected for demographic use.

All eligible subjects will be asked to fill out the Patient Health Questionnaire Depression Self-test (PHQ-9) and who score 10-19 on the PHQ-9 will be entered for a Structured Clinical Interview for Hamilton Rating Scale for Depression (HAMD). This interview will be conducted in person by our psychiatrist Dr. Chan Wai-Chi from Department of Psychiatry, the University of Hong Kong in Queen Mary Hospital. They will be divided into 2 groups by randomization. (Group A n=18, Group B n=18) The participants will receive 2 acupuncture session per week for 3 consecutively weeks. In each treatment session, all subjects in both groups will receive the same amount of needle insertion ( total 14 needles) , all needles will be retained for 30 minutes. The whole treatment will last for around 45 minutes. No sedation will be conducted.

Subjects in Group A will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation", all needles will be retained for 30 minutes. Acupoint combination: Taichong太衝 (LR 3), Ligou蠡沟 (LR 5), Zhongdu 中都(LR6), Xiguan膝關 (LR 7), Ququan曲泉 (LR 8), Zhangmen章門(LR13), Qimen期門 (LR14).

Subjects in Group B will receive 14 needles based on the TCM theory "Soothing liver-qi stagnation" and "Tonifying the heart and the spleen"and "Invigorating the Yang Qi", all needles will be retained for 30 minutes. Acupoint combination: Taichong太衝 (LR 3), , Sanyinjiao 三陰交 (SP 6), Xuanzhong懸鐘 (GB 39), Shenmen 神門 (HT 7), Zusanli 足三里(ST 36), Baihui 百會(DU 20), Shenting神庭(DU24), Qihai 氣海(RN6), Guanyuan 關元(RN4). Teding Diancibo Pu (abbreviation: TDP) "特定電磁波譜" will be applied to Group B immediately after the needle insertion. This TDP device is a infra-red heat lamp which is commonly used by acupuncturists and Chinese Medicine Practitioner as a therapeutic substitute for moxibustion. The procedure will be lasted for 30 minutes in 30-40 cm above the specified acupoint Qihai 氣海(RN6) and Guanyuan 關元(RN4).

Skin around these points will be sterilized by 75% alcohol and then sterilized disposable needle will be inserted at each point. A registered Chinese medicine practitioner with at least 5 years experience will be recruited to deliver the acupuncture treatment. The acupuncture treatment will be conducted in either Specialist Clinical Centre for Teaching and Research of School of Chinese Medicine, the University of Hong Kong (Address: G/F, 10 Sassoon Road, Pokfulam, Hong Kong), or The Hong Kong Tuberculosis Association Chinese Medicine Clinic cum Training Centre of the University of Hong Kong (Address: 2/F Tang Shiu Kin Hospital, 282 Queen's Road East, Wanchai, HK)

During the study period, subjects can receive the routine western treatment.

fNIRS will be conducted during the whole procedure of the treatment in the 1st treatment sessions and the last treatment session (6th treatment). This is a safe and non-invasive imaging to assess the brain activation. Brain activation hemodynamic signals (e.g., concentration level of Oxygenated Hemoglobin (O2Hb) and Deoxygenated Hemoglobin (HHb)) over the left dorsolateral prefrontal cortex (DLPFC) will be measured by a customized portal fNIRS device.

Subjects will be required to fill in a Patient Health Questionnaire (PHQ-9) at the following time point:

1. Screening stage
2. Before start of 1st treatment in Week 1
3. Immediately after the 3rd treatment in Week 2
4. 1st week, 2nd week and 4th week after the last treatment, conducted by telephone

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65;
2. Primary diagnosis as moderate and moderate severe depression;
3. Patient Health Questionnaire Depression Self-test (PHQ-9) score 10-19.

Exclusion Criteria:

1. Patients with primary diagnosis as Major Depressive Disorder, any history of psychosis or mania.
2. Conditions that may make it difficult to conclusively determine that depressive symptoms are the result of Depression and not some other condition: any form of substance abuse or dependence within the last 6 months, relevant medical conditions that may be the medical basis of a depression including epilepsy, history of an abnormal EEG, severe head trauma, or stroke.
3. Serious uncontrolled medical conditions [e.g. poorly controlled diabetes, severe congestive heart failure], or other medical conditions that have not been stable for at least 3 months;
4. Received Electroconvulsive therapy (ECT) in the past year.
5. Current active suicidal or self-injurious potential necessitating immediate treatment
6. Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change of Brain activation hemodynamic signals in 6 acupuncture sessions (concentration level of Oxygenated Hemoglobin (O2Hb) over the left dorsolateral prefrontal cortex (DLPFC) | 5 minutes before, during and 10 minutes after the 1st and the last (6th) acupuncture treatment session.
  Will be measured by a customized portal fNIRS device
Change of Brain activation hemodynamic signals in 6 acupuncture sessions (Deoxygenated Hemoglobin (HHb)) over the left dorsolateral prefrontal cortex (DLPFC) | 5 minutes before, during and 10 minutes after the 1st and the last (6th) acupuncture treatment session.
  Will be measured by a customized portal fNIRS device

SECONDARY OUTCOMES:
PHQ-9 | 1. Screening stage; 2. Before start of 1st treatment in Week 1; 3. Immediately after the 2nd treatment in Week 3;4. 1st week, 2nd week and 4th week after the last treatment, conducted by telephone

CONTACTS AND LOCATIONS:
Overall Officials: Jun mei Wu, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Chinese Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No